CLINICAL TRIAL: NCT03593629
Title: HIV Self-Testing to Improve the Efficiency of PrEP Delivery
Brief Title: Kenya HIV Self-Testing in PrEP Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jared Baeten, Professor, School of Medicine: Global Health; Dept. of Medicine, Allergy & Infectious Diseases, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003750; 1R01MH113572 (NIH)
Record Dates: First submitted 2018-06-02; First posted 2018-07-20 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: HIV-1-infection
Keywords: HIV; AIDS; PrEP; Truvada; Public Health; Global Health; Infectious Disease; Self-Testing; Kenya; Africa; Low and/or Middle Income Countries (LMIC); Cost-Effectiveness
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (No Intervention): Participants receive standard of care for PrEP, including 3-months of PrEP supply and HIV testing at clinic every three months
- Blood-based HIV self-testing (Experimental): Participants receive 6-months of PrEP supply and blood-based HIV self-tests for quarterly HIV testing.
  Interventions: Combination Product: 6-month PrEP + blood-based HIV self-test
- Oral fluid HIV self-testing (Experimental): Participants receive 6-months of PrEP supply and oral fluid HIV self-tests for quarterly HIV testing.
  Interventions: Combination Product: 6-month PrEP + oral fluid HIV self-test

INTERVENTIONS:
Combination Product: 6-month PrEP + blood-based HIV self-test — Participants receive 6-month PrEP supply plus two blood-based HIV self-tests (Atomo Diagnostics Blood-Based HIV-1 Self-Testing Kit) for quarterly HIV testing.
  Arms: Blood-based HIV self-testing
Combination Product: 6-month PrEP + oral fluid HIV self-test — Participants receive 6-month PrEP supply plus two oral fluid HIV self-tests (OraQuick Oral Fluid-based HIV-1 Self-Testing Kit) for quarterly HIV testing.
  Arms: Oral fluid HIV self-testing

SUMMARY:
In a three-arm, randomized trial, the investigators will test the use of HIV-1 self-testing to decrease the frequency and burden of clinic visits for PrEP while resulting in equivalent PrEP adherence and HIV testing.

DETAILED DESCRIPTION:
Guidelines recommend HIV-1 testing quarterly for individuals on PrEP. Clinic-based HIV testing every three months is costly for both clinics and participants. The investigators propose using HIV self-testing to replace quarterly clinic-based HIV testing for participants on PrEP, eliminating half of clinic visits and saving staffing and participant costs. The investigators want to understand the effect that reduced clinic contact frequency (resulting from HIV self-testing) has on PrEP adherence or completion of HIV-1 testing, overall and in subgroups.

The investigators will enroll roughly 495 eligible individuals on PrEP: 165 men and 165 women in HIV-1 serodiscordant couples and 165 women at risk of HIV-1 infection (priority populations for PrEP delivery in Kenya and more generally in Africa).

In this study, participants will be randomly assigned in a 2:1 fashion to either six-monthly clinic visits or quarterly clinic visits. Participants randomized to six-monthly clinic visits will receive a 6-month supply of PrEP and either two blood-based HIV self-tests (blood-based HIV self-testing arm) or two oral fluid HIV self-tests (oral fluid HIV self-testing arm). Participants randomized to quarterly clinic visits will receive a 3-month supply of PrEP and get tested for HIV by a healthcare professional at the clinic (standard of care arm)

Study outcomes, measured at Months 6 and 12, include PrEP adherence (defined as the detection of PrEP in dried blood spots as well as persistence in refilling PrEP), HIV-1 testing, and safety (including side effects and social harm).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years HIV-1 uninfected based on negative HIV-1 rapid testing
* Not currently enrolled in an HIV-1 prevention clinical trial
* Taking PrEP and planning to continue
* Willing to be randomized to either clinic based HIV-1 testing or HIV-1 self-testing
* Note: Women who are pregnant at screening/enrollment are still eligible

Exclusion Criteria:

* Unable to provide written informed consent
* Contraindication to use Tenofovir (TDF)+/- Emtricitabine (FTC)/ Lamivudine (3TC)

For the HIV-1 serodiscordant couples, HIV-1 infected members of the couple will be enrolled for a single visit at baseline, if:

* Age ≥18
* Able and willing to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 790 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Baeten, MD, PhD, Principal Investigator — University of Washington; Kenneth Ngure, PhD, MPH, Principal Investigator — Jomo Kenyatta University of Agriculture and Technology
Locations (1):
- Partners in Health Research and Development - Thika House, Thika, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangale DI, Heitner J, Ortblad KF, Mogere P, Kiptinness C, Mugo NR, Baeten JM, Ngure K, Barnabas R. Opportunity for cost savings with a novel differentiated model of PrEP delivery: a comparative costing analysis of six-month PrEP supported by interim HIV self-testing and standard of care PrEP dispensing in Kenya. BMC Health Serv Res. 2025 Jul 1;25(1):865. doi: 10.1186/s12913-025-12891-7. PMID 40598383
- [Derived] Thuo N, Bardon AR, Mogere P, Kiptinness C, Casmir E, Wairimu N, Owidi E, Okello P, Mugo NR, Baeten JM, Ngure K, Ortblad KF. Acceptability of six-monthly PrEP dispensing supported with interim HIV self-testing to simplify PrEP delivery in Kenya: findings from qualitative research. BMC Health Serv Res. 2024 Oct 24;24(1):1281. doi: 10.1186/s12913-024-11521-y. PMID 39448999
- [Derived] Ortblad KF, Bardon AR, Mogere P, Kiptinness C, Gakuo S, Mbaire S, Thomas KK, Mugo NR, Baeten JM, Ngure K. Effect of 6-Month HIV Preexposure Prophylaxis Dispensing With Interim Self-testing on Preexposure Prophylaxis Continuation at 12 Months: A Randomized Noninferiority Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2318590. doi: 10.1001/jamanetworkopen.2023.18590. PMID 37318803
- [Derived] Ngure K, Ortblad KF, Mogere P, Bardon AR, Thomas KK, Mangale D, Kiptinness C, Gakuo S, Mbaire S, Nyokabi J, Mugo NR, Baeten JM. Efficiency of 6-month PrEP dispensing with HIV self-testing in Kenya: an open-label, randomised, non-inferiority, implementation trial. Lancet HIV. 2022 Jul;9(7):e464-e473. doi: 10.1016/S2352-3018(22)00126-6. PMID 35777410
- [Derived] Ortblad KF, Kearney JE, Mugwanya K, Irungu EM, Haberer JE, Barnabas RV, Donnell D, Mugo NR, Baeten JM, Ngure K. HIV-1 self-testing to improve the efficiency of pre-exposure prophylaxis delivery: a randomized trial in Kenya. Trials. 2019 Jul 4;20(1):396. doi: 10.1186/s13063-019-3521-2. PMID 31272495

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-positive Partners: Participants receive a baseline questionnaire, there are no outcomes related to this group.
Period: Overall Study
Arm/Group | Standard of Care | Blood-based HIV Self-testing | HIV-positive Partners | Oral Fluid HIV Self-testing
Started | 166 | 166 | 291 | 163
Completed | 166 | 166 | 291 | 163
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HIV- Positive Partners: Participants receive a baseline questionnaire, there are no outcomes related to this group.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Blood-based HIV Self-testing | Oral Fluid HIV Self-testing | HIV- Positive Partners | Total
Number analyzed (Participants) | 166 | 166 | 163 | 291 | 786
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 2 | 1 | 7
  Between 18 and 65 years | 163 | 164 | 161 | 290 | 778
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [28 to 40] | 32 [27 to 39] | 33 [28 to 40] | 35 [28 to 43] | 33 [28 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 56 | 54 | 130 | 295
  Male | 111 | 110 | 109 | 161 | 491
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 166 | 166 | 163 | 291 | 495

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adherence to PrEP at 6 Months
Description: Laboratory tests will be conducted to measure adherence to PrEP medication by testing drug levels in the collected blood specimen. The detection of PrEP in blood will be considered as adherent to PrEP.
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Blood-based HIV Self-testing | Oral Fluid HIV Self-testing
Number analyzed (Participants) | 166 | 166 | 163
Participants | 95 | 106 | 94
Statistical Analysis 1: Comparison: Standard of Care; Test type: Non-Inferiority — Non-inferiority margin was defined as -10%; Risk Difference (RD) = 2.37, 95% CI 1-sided [lower limit -5.05]

2. Primary Outcome: Persistence in Refilling PrEP
Description: The percentage of participants that return to clinic to refill their PrEP medication. An alternative measure of PrEP adherence.
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Blood-based HIV Self-testing | Oral Fluid HIV Self-testing
Number analyzed (Participants) | 166 | 166 | 163
Participants | 134 | 127 | 130
Statistical Analysis 1: Comparison: Standard of Care vs Blood-based HIV Self-testing vs Oral Fluid HIV Self-testing; Test type: Non-Inferiority — non-inferiority margin is defined as -10%; Risk Difference (RD) = -2.60, 95% CI 1-sided [lower limit -8.88]

3. Primary Outcome: HIV-1 Testing
Description: Self-reported HIV-1 testing in the past 6 months
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Blood-based HIV Self-testing | Oral Fluid HIV Self-testing
Number analyzed (Participants) | 166 | 166 | 163
Participants | 140 | 135 | 139
Statistical Analysis 1: Comparison: Standard of Care vs Blood-based HIV Self-testing vs Oral Fluid HIV Self-testing; Test type: Non-Inferiority — non-inferiority margin is defined as -10%; Risk Difference (RD) = -1.15, 95% CI 1-sided [lower limit -6.89]

4. Secondary Outcome: PrEP Adherence
Description: as for outcome 1
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

5. Secondary Outcome: Persistence in Refilling PrEP
Description: as for outcome 2
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

6. Secondary Outcome: HIV-1 Testing
Description: Self-reported HIV-1 testing in the past 6 months
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

7. Other Pre Specified Outcome: Recent Abuse by a Sexual Partner
Description: Self-reported verbal, physical or emotional abuse by a sexual partner
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

8. Other Pre Specified Outcome: Recent Abuse by a Sexual Partner
Description: Self-reported verbal, physical or emotional abuse by a sexual partner
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

9. Other Pre Specified Outcome: Prevalence of Depression
Description: The Patient Health Questionnaire-9 item (PHQ-9) depression scale. A 0-27 point scale where scores 10 or greater can be categorized as likely depression.
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

10. Other Pre Specified Outcome: Prevalence of Depression
Description: as for outcome 9
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

11. Other Pre Specified Outcome: Participant's Self-reported Self-efficacy
Description: Measured using the General Self-Efficacy Scale (GSE), which is correlated to emotion, optimism, work satisfaction, to measure self-efficacy. The scale ranges from 10-40 points - higher scores indicate more self-efficacy.
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

12. Other Pre Specified Outcome: Participant's Self-reported Self-efficacy
Description: as for outcome 11
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

13. Other Pre Specified Outcome: Number of Sexual Partners
Description: Self-reported number of sexual partners in the past month
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

14. Other Pre Specified Outcome: Number of Sexual Partners
Description: Self-reported number of sexual partners in the past month
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

15. Other Pre Specified Outcome: Inconsistent Condom Use
Description: Participants were asked how many times they had sexual intercourse in the past month and how many times a condom was used. If condoms were not used at every time, condom use was categorized as inconsistent.
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

16. Other Pre Specified Outcome: Inconsistent Condom Use
Description: as for outcome 15
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

17. Other Pre Specified Outcome: PrEP Disclosure
Description: Participants report that at least one other person (besides one's main sexual partners in serodiscordant couples) is aware they are taking PrEP.
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

18. Other Pre Specified Outcome: PrEP Disclosure
Description: as for outcome 17
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

19. Other Pre Specified Outcome: HIV Testing Preferences
Description: Participants report their preference for HIV testing from the following options: blood-based HIV self-testing, oral HIV self-testing, testing for HIV at a standard healthcare facility
Time Frame: Month 6
Reporting Status: Not Posted, anticipated posting 2024-10

20. Other Pre Specified Outcome: HIV Testing Preferences
Description: as for outcome 19
Time Frame: Month 12
Reporting Status: Not Posted, anticipated posting 2024-10

21. Other Pre Specified Outcome: Number of Participants That Test HIV-1 Positive Since Trial Enrollment
Description: The proportion of participants (binary outcome) that test HIV-1 positive since trial enrollment. Genotypic HIV-1 resistance for seroconverters will additionally be measured.
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Blood-based HIV Self-testing | Oral Fluid HIV Self-testing
Number analyzed (Participants) | 166 | 166 | 163
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Standard of Care | Blood-based HIV Self-testing | HIV-positive Partners | Oral Fluid HIV Self-testing
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/166 | 0/291 | 0/163
Serious Adverse Events (participants affected / at risk) | 1/166 | 2/166 | 0/291 | 2/163
Other Adverse Events (participants affected / at risk) | 0/166 | 0/166 | 0/291 | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (N=166) | Blood-based HIV Self-testing (N=166) | HIV-positive Partners (N=291) | Oral Fluid HIV Self-testing (N=163)
Hospitalization, hysterectomy (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 — Hysterectomy, dysfunctional uterine bleeding; unrelated to study medication
Hospitalization, Intrauterine fetal death (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Hospitalization and induced delivery due to Intrauterine fetal death ; unrelated to study medication
Hospitalization, caesarian (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 — Caesarian section; unrelated to study medication
Hospitalization, normal delivery (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 — Normal delivery; unrelated to study medication
Hospitalization, ectopic pregnancy (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 — Ectopic pregnancy; unrelated to study medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03593629/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/29/NCT03593629/SAP_001.pdf